CLINICAL TRIAL: NCT05545852
Title: A Multicenter, Randomized, Controlled Clinical Study on the Feasibility and Safety of Gasless Transaxillary Posterior Endoscopic and Open Thyroidectomy for Papillary Thyroid Cancer.
Brief Title: A Clinical Study of Transaxillary Endoscopic and Open Thyroidectomy for PTC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-2021-324
Record Dates: First submitted 2022-08-29; First posted 2022-09-19 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Papillary Thyroid Cancer
Keywords: endoscopic; thyroidectomy
MeSH Terms: conditions — Thyroid Cancer, Papillary

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): Gasless Transaxillary Posterial Endoscopic Thyroidectomy and Ipsilateral Central Lymph Node Dissection
  Interventions: Procedure: GTPET(Gasless Transaxillary Posterial Endoscopic Thyroidectomy)
- Control Group (Active Comparator): Conventional Open Thyroidectomy and Ipsilateral Central Lymph Node Dissection
  Interventions: Procedure: COT(Conventional Open Thyroidectomy)

INTERVENTIONS:
Procedure: GTPET(Gasless Transaxillary Posterial Endoscopic Thyroidectomy) — Gasless Transaxillary Posterial Endoscopic Thyroidectomy and Ipsilateral Central Lymph Node Dissection
  Arms: Study Group
Procedure: COT(Conventional Open Thyroidectomy) — Conventional Open Thyroidectomy and Ipsilateral Central Lymph Node Dissection
  Arms: Control Group

SUMMARY:
To evaluate the feasibility and safety of gasless transaxillary posterior endoscopic thyroidectomy (Resection of thyroid lobe and isthmus, lymph node dissection in the central area of the affected side) and open radical thyroidectomy (Resection of thyroid lobe and isthmus, lymph node dissection in the central area of the affected side) as the current standard surgical treatment mode in terms of feasibility and safety of radical thyroidectomy.

DETAILED DESCRIPTION:
Subjects that suffering from papillary thyroid carcinoma will be randomized into Study Group (gasless transaxillary posterior endoscopic thyroidectomy ) or Control Group (conventional open thyroidectomy). Measure the outcomes as following, early complication rate, life quality score, the number of dissected lymph nodes, the volume of residual gland, 3-year recurrence rate, operation duration, hospital stays, hospitalization expense, and inflammatory and immune response.

ELIGIBILITY:
Inclusion Criteria:

* The patient's informed consent;
* 18 years old < age < 70 years old;
* Papillary thyroid carcinoma (Bethesda grade V-VI) was pathologically diagnosed by fine needle aspiration biopsy of the primary thyroid tumor before surgery;
* Color Doppler TI-RADS 4c-5 of primary thyroid tumor;
* The preoperative clinical staging is T1, N0-1a, M0 (see diagnostic criteria for details; according to AJCC-8th TNM tumor staging);
* It is expected that R0 surgical results can be obtained by performing single thyroid lobectomy and isthmus resection + ipsilateral central lymph node dissection;
* Preoperative ASA score I-III.

Exclusion Criteria:

* Pregnant or lactating patients;
* Suffering from serious mental illness;
* Preoperative imaging examinations suggest that the tumor is located in the thyroid isthmus or involves bilateral lobes;
* Preoperative imaging examinations suggest the possibility of cervical lateral lymph node or distant metastasis;
* Hashimoto's thyroiditis combined with hyperthyroidism or abnormal thyroid function;
* History of neck surgery;
* History of thyroid surgery (including ablation therapy for thyroid nodules);
* Family history of thyroid cancer;
* History of childhood ionizing radiation exposure;
* History of other malignant diseases within 5 years;
* A history of unstable angina or myocardial infarction within 6 months;
* History of cerebral infarction or cerebral hemorrhage within 6 months;
* History of continuous systemic corticosteroid therapy within 1 month;
* Concurrent surgical treatment of other diseases is required;
* Patients who are judged by the investigator to be unsuitable to participate in this trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Early complication rate | 30 days after surgery
  Early complications include hemorrhage, surgical site infection, recurrent laryngeal nerve injury, hypoparathyroidism (PTH<15pg/ml, or showing hypocalcification symptoms), chyle leakage, trachea injury, esophageal injury, etc.
Life quality score (3 days after surgery) | 3 days after surgery
  Use a modified Thyroid Cancer-Specific Quality of Life Questionnaire (THYCA-QOL) to measure the quality of life 3 days after surgery.
Life quality score (1 month after surgery) | 1 month after surgery
  Use a modified Thyroid Cancer-Specific Quality of Life Questionnaire (THYCA-QOL) to measure the quality of life 1 month after surgery.
Life quality score (3 months after surgery) | 3 months after surgery
  Use a modified Thyroid Cancer-Specific Quality of Life Questionnaire (THYCA-QOL) to measure the quality of life 3 months after surgery.
Life quality score (6 months after surgery) | 6 months after surgery
  Use a modified Thyroid Cancer-Specific Quality of Life Questionnaire (THYCA-QOL) to measure the quality of life 6 months after surgery.
Life quality score (1 year after surgery) | 1 year after surgery
  Use a modified Thyroid Cancer-Specific Quality of Life Questionnaire (THYCA-QOL) to measure the quality of life 1 year after surgery.

SECONDARY OUTCOMES:
The number of dissected lymph nodes | 3 days after surgery
  Record the number of harvest and metastatic lymph nodes.
The volume of residual gland | 6 month after surgery
  Measure the volume of residual gland with ultrasound tests.
3-year recurrence rate | 3 years after surgery
  The rate will be calculated from the day of randomization to the present of evidence of recurrence.
Operation duration | Intraoperative
  Record the time from skin discission to incision close.
Hospital stays | 3 days after surgery
  Record the days from the day of surgery to the day of discharge.
Hospitalization expense | 3 days after surgery
  The total hospitalization expense.
Inflammatory response | 1 day after surgery
  Examine the white blood cell count (WBC), neutrophil count (NEU) and c-reactive protein (CRP) 1 day after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Shangtong Lei, Dr., Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong, China

REFERENCES:
- See also: Registration on Chinese Clinical Trial Registry — http://www.chictr.org.cn/showproj.aspx?proj=51290